CLINICAL TRIAL: NCT00340080
Title: A Phase IV, Randomised, Multicentre, Double-blind, Study to Evaluate the Clinical Utility of Prospective Genetic Screening (HLA-B*5701) for Susceptibility to Abacavir Hypersensitivity
Brief Title: Clinical Utility Of Genetic Screening For HLA-B*5701, On Susceptibility To Abacavir Hypersensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNA106030; PREDICT-1
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infection
Keywords: Abacavir; Pharmacogenetics; hypersensitivity; HLA-B*5701
MeSH Terms: conditions — HIV Infections; Hypersensitivity | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir

SUMMARY:
Study to evaluate the utility of prospective HLA-B*5701 screening on the incidence of abacavir hypersensitivity (ABC HSR) in 1800 previously ABC-naive adults with HIV-1 from Europe, Australia and other countries as applicable. The study has two (co-primary) objectives: i) to determine if screening for HLA-B*5701 prior to ABC-containing HAART results in a lower incidence of clinically-suspected HSR versus current standard of care (no genetic screening) and ii) to determine if screening for HLA-B*5701 prior to ABC-containing HAART, results in a significantly lower incidence of immunologically-confirmed HSR versus current standard of care (no genetic screening or patch testing). The study consists of up to a 28-day screening period, a randomised observation period (Day 1 through Week 6) and, for subjects experiencing a suspected ABC HSR and a subset of ABC-tolerant subjects, an epicutaneous patch test (EPT) assessment period. Eligible subjects will be randomised to one of two study arms: a Current Standard of Care Arm (no prospective genetic screening: Control) and a Genetic Screening Arm (prospective genetic screening). Subjects identified as HLA-B*5701 positive in the prospective Genetic Screening Arm will not receive ABC and will be excluded from further study. Subjects who experience suspected ABC HSR during the 6-week observation will be withdrawn from ABC-containing product and undergo EPT patch testing 6 weeks later.

ELIGIBILITY:
Inclusion criteria:

* Infected with documented HIV-1.
* Subjects are Abacavir-naive (subjects can be antiretroviral therapy (ART)-naive or experienced).
* All subjects must have a clinical need for treatment with Abacavir (ABC) or an ABC-containing product that precedes the decision to participate in the study.
* If subjects are therapy naive they must meet the criteria for commencing HAART according to local guidelines.
* ABC and ABC-containing products are not recommended during pregnancy. A female is eligible to enter and participate in the study if she is of:

  1. Non-child-bearing potential: women who are surgically sterile or post-menopausal, the latter indicated by history of no menses for a minimum of 1 year from the date of the screening visit.
  2. Child-bearing potential: women who provide a negative pregnancy test (beta-human chorionic gonadotrophin; beta-HCG) at Screening and who agree to one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the approved product label and the instructions of a physician, during the study period and through epicutaneous patch testing where appropriate):
* Complete abstinence from intercourse from 4 weeks prior to administration of the ABC-containing compound, throughout the study, and for at least 4 weeks after discontinuation of ABC or ABC-containing product.
* Double barrier method (e.g., male condom/spermicide, male condom/diaphragm, diaphragm/spermicide). Hormonal contraceptives will not be considered sufficient forms of contraception for this study.
* Any intrauterine device with published data showing that the expected failure rate is <1% per year.
* Sterilisation (male partner of female subject).

Exclusion criteria:

* Has previously received ABC-containing therapy.
* Satisfies any contraindications or restrictions to ABC therapy as listed in the product labels. Treatment with ABC must be in line with the recommendations of the product label.
* The subject or any of their healthcare providers is aware of the subjects HLA type.
* Has undergone an allogeneic bone marrow transplant.
* Has an active or acute CDC Clinical Category C event at screening. Treatment for the acute event must have been completed at least 30 days prior to Screening.
* Current severe illness, including liver and renal failure, major organ allograft, malignancy requiring parenteral chemotherapy that can not be discontinued for the duration of the trial, or any other conditions which, in the opinion of the Investigator, would make the patient unsuitable for the study.
* Any laboratory abnormality at Screening which, in the opinion of the Investigator, should preclude the subject's participation in the study.
* Pregnant women or women who are breastfeeding.
* Any immunisation within 30 days prior to Day 1.
* Subject is, in the opinion of the Investigator, unable to complete the 6 week Observation period and the EPT assessments as required.
* Subject requires treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to Screening, or has an anticipated need for these agents within the study period.
* Subject is enrolled in one or more investigational drug/vaccine protocols.
* In France, an eligible subject is neither affiliated with nor a beneficiary of a social security category.
* A subject will not be eligible for progression to Baseline (Day 1) if any of the following criteria apply:
* A positive result for HLA-B*5701 in those subjects randomised to the genetic screening arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1806
Dates: Start 2006-04

PRIMARY OUTCOMES:
Incidence of clinically-suspected ABC HSR during the 6-week observation period. Incidence of immunologically-confirmed ABC HSR. The clinical diagnosis of which occurs over the 6-week observation period.

SECONDARY OUTCOMES:
Incidence of clinically-suspected ABC HSR in Caucasians and in different ethnic sub-groups. Sensitivity and specificity, positive and negative predictive value of genetic screening for HLA-B*5701 for susceptibility of HSR.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MB BS MRCP FFPM, Study Director — GlaxoSmithKline
Locations (211):
- Australia (2):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Miami, Queensland
- Austria (5):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- France (50):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Fréjus
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Niort
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Quimper
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Brieuc
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Germain-en-Laye
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Troyes
  - GSK Investigational Site, Valence
  - GSK Investigational Site, Valenciennes
  - GSK Investigational Site, Villejuif
- Germany (21):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Dublin, Ireland
- Israel (4):
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (29):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Latina, Lazio
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sanremo (im), Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Busto Arsizio (va), Lombardy
  - GSK Investigational Site, Cuggiono (mi), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Asti, Piedmont
  - GSK Investigational Site, Pallanza (Verbania), Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Torrette Di Ancona (an), The Marches
  - GSK Investigational Site, Bolzano, Trentino-Alto Adige
  - GSK Investigational Site, Grosseto, Tuscany
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Treviso, Veneto
  - GSK Investigational Site, Vicenza, Veneto
- GSK Investigational Site, Riga, Latvia
- Netherlands (11):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Flushing
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Zwolle
- Norway (2):
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Oslo
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- Portugal (8):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Aveiro
  - GSK Investigational Site, Cascais
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Monte Funchal
  - GSK Investigational Site, Ponta Delgada
  - GSK Investigational Site, Porto
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Iași
- Russia (15):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, N.Novgorod
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Volgograd
- GSK Investigational Site, Ljubljana, Slovenia
- Spain (24):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Calella
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Reus
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Tarragona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo ( Pontevedra)
  - GSK Investigational Site, Vitoria-Gasteiz
- Switzerland (7):
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bruderholz
  - GSK Investigational Site, La Chaux-de-Fonds
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich
- United Kingdom (18):
  - GSK Investigational Site, Derby, Derbyshire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Stoke-on-Trent, Staffordshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Dudley, Birmingham
  - GSK Investigational Site, East Yorkshire
  - GSK Investigational Site, Farnworth, Bolton
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Plaistow, London
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Derived] Mallal S, Phillips E, Carosi G, Molina JM, Workman C, Tomazic J, Jagel-Guedes E, Rugina S, Kozyrev O, Cid JF, Hay P, Nolan D, Hughes S, Hughes A, Ryan S, Fitch N, Thorborn D, Benbow A; PREDICT-1 Study Team. HLA-B*5701 screening for hypersensitivity to abacavir. N Engl J Med. 2008 Feb 7;358(6):568-79. doi: 10.1056/NEJMoa0706135. PMID 18256392